CLINICAL TRIAL: NCT02413697
Title: A Randomised Control Trial of Three-dimensional Versus Two-dimensional Ultrasound Guided Embryo Transfer in Women Undergoing Artificial Reproductive Technology Treatment
Brief Title: Three-dimensional Versus Two-dimensional Ultrasound Guided Embryo Transfer in Women Undergoing ART Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Sotirios Saravelos, Dr, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRE-2014.650
Record Dates: First submitted 2015-04-04; First posted 2015-04-10 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Two-dimensional ultrasound (Active Comparator): Two-dimensional ultrasound guided embryo transfer
  Interventions: Device: Two-dimensional ultrasound
- Three-dimensional ultrasound (Experimental): Three-dimensional ultrasound guided embryo transfer
  Interventions: Device: Three-dimensional ultrasound

INTERVENTIONS:
Device: Two-dimensional ultrasound — Two-dimensional ultrasound guided embryo transfer
  Arms: Two-dimensional ultrasound
Device: Three-dimensional ultrasound — Three-dimensional ultrasound guided embryo transfer
  Arms: Three-dimensional ultrasound

SUMMARY:
Objectives: To assess whether embryo transfer guided by three-dimensional ultrasound (3DUS) produces a significantly higher clinical pregnancy rate than embryo transfer guided by two-dimensional ultrasound (2DUS).

Hypothesis: 3DUS guided embryo transfer will produce a significantly higher clinical pregnancy rate compared with 2DUS guided embryo transfer. Design and subjects: Prospective randomised control trial (RCT) at the Prince of Wales Hospital. Inclusion criteria include women undergoing embryo transfer in fresh and frozen cycles. Exclusion criteria include women aged >42 years and women whose endometrial cavity cannot be visualised adequately via US. Power calculations indicate that 232 patients per arm are required to demonstrate an increase of 12% in clinical pregnancy rates.

Study instruments: US examinations will be performed using a General Electric(GE) Voluson series US machine with a standard 3D transvaginal probe. For embryo transfer, the Cooks Guardia Access EchoTip catheter will be used.

Interventions: 3D versus 2DUS for guidance during embryo transfer. Main outcome measures: clinical pregnancy. Secondary outcome measures: implantation rate, multiple pregnancy, miscarriage, ectopic pregnancy and live birth rates.

Data analysis: Data processing and analysis will be performed using the Statistical Packages of Social Sciences for Windows (SPSS, Inc). Descriptive and comparative statistical methods will be used to analyse the primary outcomes. P-values of <0.05 will be considered significant.

Expected results: The study arm undergoing 3DUS guided embryo transfer are expected to have an improved clinical pregnancy rate compared with the control arm undergoing 2DUS guided embryo transfer.

DETAILED DESCRIPTION:
INTRODUCTION

The role and use of 2DUS in gynaecology is undisputed as it forms an integral part of diagnosing pathologies of the uterus, tubes and ovaries. In reproductive medicine, it is of particular significance as it is additionally the most widespread tool available to monitor endometrial thickness, follicular status and growth, allow guided retrieval of oocytes from the ovary and also guided transfer of fertilised embryos into the uterus [1]. These are undoubtedly some of the most critical procedures/steps of ART.

The development of 3DUS has brought somewhat of a breakthrough in the field as now 3D volumes of images can be acquired and analysed live or retrospectively. From a practical perspective, the scanning procedure does not differ from the routine 2D US and the acquisition of a 3D volume requires only a few seconds. Analysis of these volumes allows reconstruction of planes which are not always possible with 2DUS (such as the 3D coronal plane of the uterus). As a result, 3DUS is now considered to be the most accurate non-invasive modality to diagnose uterine anomalies [2, 3]. Furthermore, 3DUS allows accurate volume calculations of structures such as the endometrium and follicles. These new possibilities, coupled with advanced software now also allows for automated measurements of these variables, which may improve accuracy, reduce interobserver variability and increase efficiency of an ART unit [4].

Several publications now in the literature support that 3DUS may play a major role in ART in the future [5-8]. Areas which 3D US may provide additional information are:

* Assessment of ovarian blood flow, follicular volume and growth [9]
* Assessment of endometrial and subendometrial blood flow and volume [10, 11]
* Assessment of precise catheter placement during embryo transfers [12] The latter is perhaps the area which has been the least investigated so far, despite embryo transfer being arguably the step of highest importance throughout the entire ART process. Two preliminary studies have shown that 3DUS guided embryo transfer significantly improves catheter placement compared with 2DUS [13] and can allow for correction of up to 20% of mal-positioned catheters where 2DUS alone has been used [14]. The largest series to date, has demonstrated that by use of 3DUS, the placement of embryos can be performed in the so called maximum implantation potential point, which is where the trajectories of the fallopian tubes meet in the centre of the uterine cavity, where the endometrial thickness and blood flow is thought to be greatest [12]. However, to our knowledge, there has been no randomised controlled trial (RCT) in the literature to systematically test 3DUS versus 2DUS guided embryo transfer with respect to pregnancy outcomes. If 3DUS guided embryo transfer is confirmed to produce a higher pregnancy rate than 2DUS guided embryo transfer, it will have significant impact on the daily clinical practice of ART units worldwide.

AIMS AND HYPOTHESES

Aims To determine if 3DUS guided embryo transfer should routinely replace 2DUS guided embryo transfer.

Hypotheses 3DUS guided embryo transfer produces a higher clinical pregnancy rate compared with 2DUS guided embryo transfer

PLAN OF INVESTIGATION

Subject recruitment Women with infertility will be recruited from the Assisted Reproductive Technology Unit of the department of Obstetrics and Gynaecological, Prince of Wales Hospital. They will be given information leaflets at the beginning of their treatment cycle, and further counselled on the day of oocyte retrieval or on the day of commencement of progesterone therapy. This will allow sufficient time to consider participation in the trial and confirm their consent on the day of embryo transfer. The investigators anticipate that over 80% of subjects undergoing embryo transfer will participate.

Study design A prospective single-blinded randomized controlled trial.

Inclusion criteria:

* Women undergoing embryo transfer in either fresh or frozen cycles.
* Women whose endometrial cavity can be visualised adequately via US Exclusion criteria
* Women aged >42 years
* Women whose endometrial cavity cannot be visualised adequately via US, such as:

Large fibroids Adenomyosis BMI>35 Significant uterine retroflexion/retroversion

Power calculation The largest published series to date using 3DUS guided embryo transfers demonstrates a clinical pregnancy rate of 37% for women with an average age of 38 [12]. Our unit in 2013 achieved a clinical pregnancy rate of 25% for women in a similar age group. Assuming that 3DUS guided embryo transfer will enable our unit to increase the clinical pregnancy rate from 25% to 37 % (an increase of 12%), a power calculation using alpha of 0.05, beta of 0.2 and power of 0.80, indicates that 232 patients per arm are required. To account for a small amount of drop-outs 480 subjects in total will be recruited.

Methods 232 women per arm will be recruited as part of this prospective randomized controlled trial. The inclusion criteria will be patients with reproductive failure undergoing IVF/ICSI embryo transfer. The exclusion criteria will be (i) women aged >42 years; (ii) women whose endometrial cavity cannot be visualised adequately via US, such as large fibroids, adenomyosis; (iii) BMI>35, and (iv) significant uterine retroflexion/retroversion. At the time of embryo transfer, patients will be assigned to either of two groups: a) the 2DUS group where they will have their embryo transferred under the guidance of 2DUS, or b) the 3DUS group, where they will have their embryo transferred under the guidance of 3DUS.

Randomisation Patients will be randomised into the 3D or 2DUS groups with a 1 to 1 ratio using a computer-generated randomisation list with blocks of 10 in sealed envelopes pre-prepared by an impartial research nurse, to ensure equal distribution of subject assignment.

Procedure The use of 2DUS guidance for embryo transfer is universally standard practice. All ultrasound examinations will be performed using the GE Voluson series ultrasound machines, with a standard 3D transvaginal probe (model RIC5-9-D; 6.6 MHz central image frequency). The examination with 3DUS will be identical to the routine 2D examination including an acquisition of a 3D volume which takes a few seconds. The 3D facility is engaged by switching into the "3D" mode. A mobile sector appears and the operator identifies the "region of interest." The acquisition is then commenced and the transducer crystal then rotates through approximately 90° for less than 10 seconds. The images are shown instantly to the operator and can be stored digitally onto the hard disc attached to ultrasonography machine for subsequent analysis. For the purpose of homogeneity and to reduce operator bias, the principal applicant (SS) will perform all 3DUS examinations.

For the purpose of homogeneity and to reduce operator bias, the principal investigator (SS) will perform all 3DUS examinations. In the 3D group, the catheter position will be corrected according to the coronal plane view of the uterus on 3DUS, aiming for the maximum implantation potential point, along the midline of the uterine cavity, as previously described in the literature [12]. In the 2D group, the catheter position will be guided in the longitudinal plane by 2DUS, according to current clinical practice. The patients will be blinded to which technique is used during the embryo transfer, but will be shown a 2D/3D image of the embryo flash after the transfer is complete and after the catheter has been removed.

Outcome measures The primary outcome measure will be the clinical pregnancy rate, defined as the presence of at least one gestational sac at 6 weeks gestation. The secondary outcome measures will include implantation rate, multiple pregnancy, miscarriage, ectopic pregnancy, and live birth rates. Miscarriage will be defined as biochemical if there is no US evidence of pregnancy and clinical if there is US evidence of pregnancy. Live birth will be considered as a baby born live after 24 weeks gestation.

Data processing and analysis The researchers will ensure the confidentiality of sensitive data by minimizing the number of personnel who handles subject data. The computer data will be encrypted as required to maximize security. All paper documents will be locked in filing cabinets, and only authorized personnel could access this information.

Data processing for statistical analysis will be performed using the Statistical Packages of Social Sciences for Windows (SPSS, Inc). Data will be presented by percentage, mean and standard deviation, median and range where appropriate. Comparisons between groups will be carried out by Student T test for continuous variables, ANOVA for mean value comparisons, Chi-square/Fisher's exact test for categorical data. Stepwise logistic regression analysis may be performed as part of systematic analysis for primary outcomes. P-values of <0.05 will be considered significant.

Monitoring and interim analysis As the study is perceived to be safe and poses no additional hazard, a Data Monitoring Committee and interim analysis is not considered necessary, in accordance with the most current Food and Drug Administration (FDA) recommendation [15].

Ethical considerations US is a safe and non-invasive examination. There are no known adverse effects of routine ultrasound to the mother or the embryo. No extra pain or discomfort is associated with the 3DUS versus 2DUS and the time difference in performing the exam is minimal. Application for ethics approval has already been submitted in December 2014 and is pending final approval.

Consent All subjects will be given detailed written explanation of the study and sufficient time to consider their participation. A written consent form will be signed by the patient and retained in our confidential records.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing embryo transfer in either fresh or frozen cycles.
* Women whose endometrial cavity can be visualised adequately via US

Exclusion Criteria:

* Women aged >42 years
* Women whose endometrial cavity cannot be visualised adequately via US, such as large fibroids, adenomyosis, BMI>35, significant uterine retroflexion/retroversion

Ages: 24 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 481 (Actual)
Dates: Start 2015-04; Primary Completion 2016-04 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy | 12 months
  Clinical pregnancy rate following ART treatment

SECONDARY OUTCOMES:
Implantation | 12 months
  Implantation rate following ART treatment
Multiple pregnancy | 12 months
  Multiple pregnancy rate following ART treatment
Miscarriage | 12 months
  Miscarriage rate following ART treatment
Ectopic pregnancy | 12 months
  Ectopic pregnancy rate following ART treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sotirios Saravelos, MBBS, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Shatin, Hong Kong

REFERENCES:
- [Background] Alcazar JL, Iturra A, Sedda F, Auba M, Ajossa S, Guerriero S, Jurado M. Three-dimensional volume off-line analysis as compared to real-time ultrasound for assessing adnexal masses. Eur J Obstet Gynecol Reprod Biol. 2012 Mar;161(1):92-5. doi: 10.1016/j.ejogrb.2011.12.002. Epub 2011 Dec 22. PMID 22197306
- [Background] Bermejo C, Martinez Ten P, Cantarero R, Diaz D, Perez Pedregosa J, Barron E, Labrador E, Ruiz Lopez L. Three-dimensional ultrasound in the diagnosis of Mullerian duct anomalies and concordance with magnetic resonance imaging. Ultrasound Obstet Gynecol. 2010 May;35(5):593-601. doi: 10.1002/uog.7551. PMID 20052665
- [Background] Saravelos SH, Cocksedge KA, Li TC. Prevalence and diagnosis of congenital uterine anomalies in women with reproductive failure: a critical appraisal. Hum Reprod Update. 2008 Sep-Oct;14(5):415-29. doi: 10.1093/humupd/dmn018. Epub 2008 Jun 6. PMID 18539641
- [Background] Raine-Fenning N, Jayaprakasan K, Deb S, Clewes J, Joergner I, Dehghani Bonaki S, Johnson I. Automated follicle tracking improves measurement reliability in patients undergoing ovarian stimulation. Reprod Biomed Online. 2009 May;18(5):658-63. doi: 10.1016/s1472-6483(10)60010-7. PMID 19549444
- [Background] Raine-Fenning N, Jayaprakasan K, Chamberlain S, Devlin L, Priddle H, Johnson I. Automated measurements of follicle diameter: a chance to standardize? Fertil Steril. 2009 Apr;91(4 Suppl):1469-72. doi: 10.1016/j.fertnstert.2008.07.1719. Epub 2008 Oct 18. PMID 18930205
- [Background] Raine-Fenning N, Fleischer AC. Clarifying the role of three-dimensional transvaginal sonography in reproductive medicine: an evidenced-based appraisal. J Exp Clin Assist Reprod. 2005 Aug 11;2:10. doi: 10.1186/1743-1050-2-10. PMID 16095530
- [Background] Coyne L, Jayaprakasan K, Raine-Fenning N. 3D ultrasound in gynecology and reproductive medicine. Womens Health (Lond). 2008 Sep;4(5):501-16. doi: 10.2217/17455057.4.5.501. PMID 19072489
- [Background] Jurkovic D. Three-dimensional ultrasound in gynecology: a critical evaluation. Ultrasound Obstet Gynecol. 2002 Feb;19(2):109-17. doi: 10.1046/j.0960-7692.2001.00654.x. No abstract available. PMID 11876800
- [Background] Raine-Fenning N, Jayaprakasan K, Clewes J, Joergner I, Bonaki SD, Chamberlain S, Devlin L, Priddle H, Johnson I. SonoAVC: a novel method of automatic volume calculation. Ultrasound Obstet Gynecol. 2008 Jun;31(6):691-6. doi: 10.1002/uog.5359. PMID 18484679
- [Background] Ng EH, Chan CC, Tang OS, Yeung WS, Ho PC. The role of endometrial and subendometrial blood flows measured by three-dimensional power Doppler ultrasound in the prediction of pregnancy during IVF treatment. Hum Reprod. 2006 Jan;21(1):164-70. doi: 10.1093/humrep/dei277. Epub 2005 Aug 25. PMID 16123083
- [Background] Ng EH, Chan CC, Tang OS, Yeung WS, Ho PC. Endometrial and subendometrial vascularity is higher in pregnant patients with livebirth following ART than in those who suffer a miscarriage. Hum Reprod. 2007 Apr;22(4):1134-41. doi: 10.1093/humrep/del458. Epub 2006 Dec 5. PMID 17148577
- [Background] Gergely RZ, DeUgarte CM, Danzer H, Surrey M, Hill D, DeCherney AH. Three dimensional/four dimensional ultrasound-guided embryo transfer using the maximal implantation potential point. Fertil Steril. 2005 Aug;84(2):500-3. doi: 10.1016/j.fertnstert.2005.01.141. PMID 16084896
- [Background] Fang L, Sun Y, Su Y, Guo Y. Advantages of 3-dimensional sonography in embryo transfer. J Ultrasound Med. 2009 May;28(5):573-8. doi: 10.7863/jum.2009.28.5.573. PMID 19389895
- [Background] Letterie GS. Three-dimensional ultrasound-guided embryo transfer: a preliminary study. Am J Obstet Gynecol. 2005 Jun;192(6):1983-7; discussion 1987-8. doi: 10.1016/j.ajog.2005.02.044. PMID 15970868
- [Derived] Saravelos SH, Kong GW, Chung JP, Mak JS, Chung CH, Cheung LP, Li TC. A prospective randomized controlled trial of 3D versus 2D ultrasound-guided embryo transfer in women undergoing ART treatment. Hum Reprod. 2016 Oct;31(10):2255-60. doi: 10.1093/humrep/dew206. Epub 2016 Sep 2. PMID 27591231
- See also: 15. Food and Drug Administration. Guidance for Clinical Trial Sponsors Establishment and Operation of Clinical Trial Data Monitoring Committees — http://www.fda.gov/downloads/RegulatoryInformation/Guidances/ucm127073.pdf